CLINICAL TRIAL: NCT06990724
Title: Effectiveness Testing of a Videogame Intervention (No Baby No) to Decrease Contraception Non-use Among Adolescents: A Randomized Trial
Brief Title: Effectiveness Testing of a Videogame Intervention (No Baby No) to Decrease Contraception Non-use Among Adolescents.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-11028189; TP2AH000081 (Other Grant/Funding Number: Department of Health and Human Services)
Record Dates: First submitted 2025-05-15; First posted 2025-05-25 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Contraceptive Usage; Contraception Behavior
MeSH Terms: conditions — Contraception Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Baby No Videogame Intervention (Experimental): Participants randomized to video game intervention for 120 minutes over two sessions within two weeks.
  Interventions: Other: Videogame Intervention
- Commercial game control (Sham Comparator): Participants randomized to commercial game intervention for 120 minutes over two sessions within two weeks.
  Interventions: Other: Commercial game control

INTERVENTIONS:
Other: Videogame Intervention — No Baby No video game
  Arms: No Baby No Videogame Intervention
Other: Commercial game control — Commercial video game
  Arms: Commercial game control

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a videogame compared to an attention/time control at reducing contraceptive non-use among adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* Age15-20 at the time of enrollment
* Able to speak and read English or Spanish
* Have a smart phone (to scan QR code) or personal email account (to take screening questionnaire)

Exclusion Criteria:

* Age less than 15 or older than 20
* Unable to speak and read English or Spanish
* Do not have a smart phone or personal email account

Ages: 15 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 850 (Estimated)
Dates: Start 2025-06-11 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Change in mean frequency of participants' contraception non-use over the last 3 months. | Baseline, 3-month follow-up, 9-month follow-up.
  Change in mean frequency of how often participants had penile/vaginal sex without a condom or birth control (pregnancy prevention), as self-reported on a customized survey with multiple-choice questions adapted from the Youth Risk Behavior Survey (YRBS). Scale values range from once to five or more times, with higher scores indicating a "worse" outcome. Scores are not being reported. At baseline, 2 weeks, and 9-month follow-up participants will be asked about the prior 3 months.
Change in mean frequency of participants' contraception non-use at last sexual encounter. | Baseline, 3-month follow-up, 9-month follow-up.
  Change in mean frequency of how often participants had penile/vaginal sex without a condom or birth control (pregnancy prevention), as self-reported on a customized survey with multiple-choice questions adapted from the Youth Risk Behavior Survey (YRBS). Scale values range from once to five or more times, with higher scores indicating a "worse" outcome. Scores are not being reported. At baseline, 2 weeks, and 9-month follow-up participants will be asked about their last sexual encounter.
Change in participants' use of different types of contraception over the last 3 months. | Baseline, 3-month follow-up, 9-month follow-up.
  A change in the mean use of less effective- (withdrawal, condom with or without spermicide, spermicide alone, fertility-based awareness, diaphragm, sponge), more effective- (pill, patch, vaginal ring, injection, intrauterine device, implant), and dual method (condom + other) contraception use during sexual encounters as self-reported on a customized survey with multiple-choice questions adapted from the Youth Risk Behavior Survey (YRBS). Participants select all forms of contraception that they used, with response options also including "No method was used to prevent pregnancy or STIs". At baseline, 2 weeks, and 9-month follow-up participants will be asked about the prior 3 months
Change in participants' use of different types of contraception at last sexual encounter. | Baseline, 3-month follow-up, 9-month follow-up.
  A change in the mean use of less effective- (withdrawal, condom with or without spermicide, spermicide alone, fertility-based awareness, diaphragm, sponge), more effective- (pill, patch, vaginal ring, injection, intrauterine device, implant), and dual method (condom + other) contraception use during sexual encounters as self-reported on a customized survey with multiple-choice questions adapted from the Youth Risk Behavior Survey (YRBS). At baseline, 2 weeks, and 9-month follow-up participants will be asked about their last sexual encounter.
Change in number of participants abstaining from having sex over the last 3 months. | Baseline, 3-month follow-up, 9-month follow-up.
  A change in the number of participants who abstained from having sex as self-reported on a customized survey with multiple-choice questions adapted from the Youth Risk Behavior Survey (YRBS). At baseline, 2 weeks, and 9-month follow-up participants will be asked about the prior 3 months.
Change in the mean number of sexual encounters over the last 3 months. | Baseline, 3-month follow-up, 9-month follow-up.
  A change in the mean number of times participants had penile/vaginal sex as self-reported on a customized survey with a multiple-choice survey question adapted from the Youth Risk Behavior Survey (YRBS). At baseline, 2 weeks, and 9-month follow-up participants will be asked about the prior 3 months.
Change in the mean number of sexual partners over the last 3 months. | Baseline, 3-month follow-up, 9-month follow-up.
  A change in participants mean number of self-reported sexual partners, as reflected by their answer to a multiple-choice survey question adapted from the Youth Risk Behavior Survey (YRBS). At baseline, 2 weeks, and 9-month follow-up participants will be asked about the prior 3 months.
Change in the number of participants who use alcohol and/or take drugs before sex at last sexual encounter. | Baseline, 3-month follow-up, 9-month follow-up.
  Change in the number of participants who self-report drinking alcohol or using drugs before having sex, based on Yes/No responses to a question adapted from the Youth Risk Behavior Survey (YRBS). At baseline, 2 weeks, and 9-month follow-up participants will be asked about the last sexual encounter.
Change in the number of participants with a positive STI (Sexually Transmitted infection) test result. | Baseline, 3-month follow-up, 9-month follow-up.
  A change in the number of participants who self-report ever receiving a positive STI result on a customized survey as adapted by YRBSS Questionnaire. At baseline, 2 weeks, and 9-month follow-up participants will be asked if they have ever received a positive STI (Sexually Transmitted infection) test result.
Change in the number of participants with a positive pregnancy test result for themselves or a partner. | Baseline, 3-month follow-up, 9-month follow-up.
  A change in the number of participants who self-report ever receiving a positive pregnancy test result or report their partner ever receiving a positive pregnancy test result, as documented by a Yes/No question on a customized survey. At baseline, 2 weeks, and 9-month follow-up participants will be asked if they/their partner have ever received a positive pregnancy test result.

SECONDARY OUTCOMES:
Change in participants' intentions for contraception non-use over the next year, as indicated by participants' mean responses to a survey question. | Baseline, 3-month follow-up, 9-month follow-up.
  A change in the mean Likert-scale rating of participants on a survey item asking about their commitment to using contraception adapted from existing literature. At baseline, 2 weeks, and 9-month follow-up participants will be asked about their commitment to using contraception.
Change in participants' self-efficacy regarding condom use, as indicated by their mean rating on a survey question. | Baseline, 3-month follow-up, 9-month follow-up.
  A change in the mean 5-point Likert-scale rating (anchor points "I strongly agree" to "I strongly disagree") on a survey item by participants reflecting their degree of confidence in correctly and consistently using condoms. The survey question is adapted from existing literature. At baseline, 2 weeks, and 9-month follow-up participants will be asked about their confidence in condom usage.
Change in participants' self-efficacy regarding contraception use, as indicated by their mean ratings on a survey question. | Baseline, 3-month follow-up, 9-month follow-up.
  A change in the mean survey-item rating by participants reflecting their degree of confidence in correctly and consistently using contraception using a question adapted from existing literature. At baseline, 2 weeks, and 9-month follow-up participants will be asked about their confidence in contraception use.
Change in participants' perceptions of sexual risk (susceptibility to getting an STI), as indicated by their mean rating on a survey question. | Baseline, 3-month follow-up, 9-month follow-up.
  A change in the mean survey-item rating by participants reflecting their perceived likelihood of getting an STI, based on contraception non-use, using a question adapted from existing literature. At baseline, 2 weeks, and 9-month follow-up participants will be asked of their perceived likelihood of getting an STI.
Change in participants' perceptions of sexual risk (getting pregnant/getting a partner pregnant), as indicated by their mean rating on a survey question. | Baseline, 3-month follow-up, 9-month follow-up.
  A change in the mean survey-item rating by participants reflecting their perceived likelihood of getting pregnant (or getting a partner pregnant), based on contraception non-use, using a question adapted from existing literature. Anchor points on the 5-point Likert scale range from "I strongly agree" to "I strongly disagree". At baseline, 2 weeks, and 9-month follow-up participants will be asked about their perceived likelihood of getting pregnant/their partner pregnant if they didn't use contraception.
Change in participants' sexual knowledge, as reflected by their mean scores on a sexual knowledge questionnaire. | Baseline, 3-month follow-up, 9-month follow-up.
  A change in participants' mean scores on questionnaire items assessing their sexual knowledge (STIs, pregnancy and contraception) using questions adapted from existing literature. Sexual knowledge questionnaire items completed by participants at baseline, 2 weeks, and 9-month follow-up.
A change in the number of participants who visit a clinic to obtain contraception or to undergo sexually transmitted infection (STI) screening over the past 3 months. | Baseline, 3-month follow-up, 9-month follow-up.
  A change in the number of participants self-reporting visiting a clinic or doctor's office to discuss or get contraception or STI screening using a question adapted from existing literature. Participants reported at baseline, 2 weeks, and 9-month follow-up.
Assessment of the fidelity of program delivery based on duration of No Baby No game play. | Baseline
  Assessment of the mean duration that each participant plays the No Baby No game over two game-play sessions (Baseline and approximately 1 week follow-up), as captured by the video game.
Assessment of the fidelity of program delivery based on number of interruptions to No Baby No game play. | Baseline
  Assessment of the average number of interruptions to game play per participant (number of times participant leaves the room or has to be redirected to play the game), as hand-recorded by research assistants over two gameplay sessions (Baseline and approximately 1 week follow-up).
Assessment of the quality of No Baby No program delivery, as indicated by the average number of technological failures during the game-play experience. | Baseline
  Assessment of the average number of technological failures during No-Baby No game play (internet-, tablet- or game failures) as hand-recorded by research assistants on game-play session checklists over two game play sessions (Baseline and approximately 1 week follow-up).
Assessment of the quality of No Baby No program delivery, as measured by the average number of minutes of game play. | Baseline
  Average number of minutes of game play across each of two game-play sessions, as captured by the No Baby No video game (Baseline and approximately 1 week follow-up).
Assessment of the quality of No Baby No program delivery, as measured by the average number of game play sessions attended by participants. | Baseline
  Average number of game play sessions attended by participants out of a maximum total of two), as captured by the No Baby No video game (Baseline and approximately 1 week follow-up).
Assessment of the quality of No Baby No program receipt, as measured by participants' average satisfaction with the game-play experience. | Baseline
  Assessment of participants' average satisfaction with the No Baby No gameplay experience, as rated on a 5-Point Likert scale after each of two game-play sessions (Baseline and approximately 1 week follow-up).
Assessment of participants' responsiveness to the No Baby No video game, as measured by their average enjoyment rating for the game. | Baseline
  Assessment of participants' average response to a multiple-choice questionnaire item asking about how much they enjoyed playing the game at two gameplay sessions (Baseline and approximately 1 week follow-up). Response options to the question "I enjoyed playing the game" are on a 5-point Likert scale with anchor points of "I strongly agree" and "I strongly disagree".
Assessment of participants' responsiveness to the No Baby No video game, as measured by their average helpfulness rating for the game. | Baseline
  Assessment of participants' average response to a multiple-choice questionnaire item asking about how helpful they found the game at two gameplay sessions (Baseline and approximately 1 week follow-up). Response options to the question "I found the game helpful" are on a 5-point Likert scale with anchor points of "I strongly agree" and "I strongly disagree".
Assessment of participants' responsiveness to the No Baby No video game, as measured by their average rating of connection with the characters from the game. | Baseline
  Assessment of participants' average response to a multiple-choice questionnaire item asking about how connected they were to the characters in the game at two gameplay sessions (Baseline and approximately 1 week follow-up). Response options to the question "I felt connected to the characters in the game" are on a 5-point Likert scale with anchor points of "I strongly agree" and "I strongly disagree".
Assessment of participants' responsiveness to the No Baby No video game, as measured by their average rating of likelihood of playing the game again. | Baseline
  Assessment of participants' average response to a multiple-choice questionnaire item asking how likely they would be to play the game again, if given the choice. Question completed at two gameplay sessions (Baseline and approximately 1 week follow-up). Response options to the question "I would play the game again" are on a 5-point Likert scale with anchor points of "I strongly agree" and "I strongly disagree".
Assessment of the acceptability of the No Baby No video game to participants, as measured by their average rating of comprehension of game content. | Baseline
  Assessment of participants' average response to a multiple-choice questionnaire item asking about how easy the content of the game was to understand. Question completed at two gameplay sessions (Baseline and approximately 1 week follow-up). Response options to the question "I found the content in the game easy to understand" are on a 5-point Likert scale with anchor points of "I strongly agree" and "I strongly disagree".
Assessment of the acceptability of the No Baby No video game to participants, as measured by their average rating of the game's usefulness. | Baseline
  Assessment of participants' average response to a multiple-choice questionnaire item asking about how useful the game was in helping participants to make real-life decisions. Question completed at two gameplay sessions (Baseline and approximately 1 week follow-up). Response options to the question "I found the game useful in helping me to make decisions in real life" are on a 5-point Likert scale with anchor points of "I strongly agree" and "I strongly disagree".
Qualitative assessment of the feasibility of the program delivery protocol for the No Baby No game, as evidenced by resource sufficiency. | Baseline
  Assessment of whether the resources provided for game-play sessions were sufficient, as documented through meeting minutes from twice-weekly team meetings with research personnel facilitating No Baby No game-play sessions (at Baseline and approximately 1 week follow-up).
Qualitative assessment of facilitators and barriers to No Baby No videogame delivery (feasibility metrics). | Baseline
  Assessment of facilitators and barriers to program delivery, as documented through meeting minutes from twice-weekly team meetings with research personnel facilitating No Baby No game-play sessions (at Baseline and approximately 1 week follow-up).

CONTACTS AND LOCATIONS:
Overall Officials: Aileen Gariepy, MD, MPH, MHS, Principal Investigator — Weill Medical College of Cornell University
Locations (7):
- United States (7):
  - Sesame Flyers International Inc., Brooklyn, New York
  - El Barrio Operation Fightback, New York, New York
  - King of Kings Foundation, Queens, New York
  - New York Center for Interpersonal Development (NYCID), Staten Island, New York
  - Bronx Health Link, The Bronx, New York
  - ASPIRA, The Bronx, New York
  - Destination Tomorrow, The Bronx, New York

IPD SHARING:
Plan to Share IPD: No